CLINICAL TRIAL: NCT04625036
Title: Pilot Study on Peripheral Vascular Function in Covid-19 Patient
Brief Title: NO-mediated Vascular Function in Covid-19 Patient
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Principal Investigator, Paola Baiardi, Principal Investigator, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: ICS Maugeri 2437 CE
Record Dates: First submitted 2020-10-30; First posted 2020-11-12 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID -19; Vascular function; Endothelial function
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: COVID-19 patients: Patients, from acute care hospitals, diagnosed with COVID-19 pneumonia, with documented positive throat swab, within one month from discharge.
  Interventions: Diagnostic Test: Single passive leg movement

INTERVENTIONS:
Diagnostic Test: Single passive leg movement — The investigation consists of a non-invasive evaluation by ultrasounds performed on the common femoral artery investigating the speed of arterial blood flow [Leg Blood Flow LBF] and diameter of vessel with a dedicated ultrasound system (General Electric Medical Systems, Milwaukee, WI) using Doppler method, before and after a passive flexion-extension movement of the knee. A linear probe will be used with a frequency of 5 MHz. Using the diameter of the artery and the average volume (Vmean), the LBF will be calculated every second with the formula=Average volume*PiGreco*(vessel diameter / 2)2*60.
  The subject will be placed in a sitting position for 20 minutes before the test. The protocol consists of image acquisition for 60 seconds (basal measurement), followed by a passive flexion-extension of the knee (single passive leg movement). The knee flexion will be performed by health care personnel at a rate of 1 Hz. At the end of the movement, the recording will continue for 60 seconds.

SUMMARY:
The 2019 coronavirus-induced infection (COVID-19) has caused a pandemic that has spread worldwide. Up to date, many subjects affected by the virus report important sequelae on different organs increasing morbidity and exacerbating previous pathological conditions. Mortality is also increased in cases of comorbidities such as cardiovascular disease, hypertension and diabetes. COVID-19 infection is caused by Coronavirus-2 (SARS-CoV-2). Concerning the specific interaction of SARS-CoV-2 with the cardiovascular system, we know that this virus enters the body through the receptors for the conversion of angiotensin II (ACE2r) that are present in the lungs, heart, intestinal epithelium and vascular endothelium. This receptor's availability suggests a multi-organ involvement with a consequent multi-organ dysfunction, as found in patients affected by SARS-CoV-2 infection.

Furthermore, poor vascular peripheral function -usually correlated with old age and long periods of bed rest or hypomobility- is a distinguishing characteristic of the population affected by COVID-19, as well. Thus, it is reasonable to expect that peripheral vascular function, already deteriorated by aging and common age-related diseases, can be further compromised by COVID-19 and by the forced hypomobility, typically experienced during the acute phase of the disease.

The main aim of this project will be to investigate the peripheral NO-mediated vascular function in the leg of patients recovering from Covid-19 pneumonia.

A significant vascular dysfunction is expected to be found in post COVID individuals and to be correlated to the relevant clinical variables.

DETAILED DESCRIPTION:
The 2019 coronavirus-induced infection (COVID-19) has caused a pandemic that has spread worldwide, causing approximately 250,000 deaths to date. Even if the contagion curves seem to stabilize, many subjects have been affected by the virus and report important sequelae on the cardiovascular system. This can be explained by the assumption that COVID-19 interacts with the cardiovascular system at different levels, increasing morbidity and exacerbating previous pathological conditions. Mortality is, in fact, increased in cases of comorbidities such as cardiovascular disease, hypertension and diabetes.

COVID-19 infection is caused by Coronavirus-2 (SARS-CoV-2). This virus enters the body through the receptor for the conversion of angiotensin [angiotensin-converting enzyme 2, ACE2]. This receptor is present in the lungs, heart, intestinal epithelium and vascular endothelium. The receptor's availability suggests a multi-organ dysfunction, as found in patients affected by SARS-CoV-2 infection. In particular, the infection of endothelial cells or pericytes, as well as the cytokine-mediated inflammatory cascade induced by the infection, can lead to severe microvascular and macrovascular dysfunctions.

It is important to underline that endothelial damage is one of the precursors of the atherosclerosis and endothelial dysfunction is related to pulmonary, cardiac and neurological diseases. Furthermore, poor vascular function is related to old age and long periods of bed rest or hypomobility, those characteristics are present in the population affected by COVID-19, as well. Thus, it is reasonable to expect that peripheral vascular function, already deteriorated by aging and common age-related diseases, can be further compromised by COVID-19 and by the forced hypomobility typically experienced during the acute phase of the disease.

Recently, the endothelial function mediated by nitric oxide (NO) has been easily and non-invasively investigated on common femoral artery with the ultrasound technique of Single Passive Leg Movement. The main aim of this project will be to investigate the NO-mediated vascular function in patients recovering from Covid-19 pneumonia, within one month from discharge in order to verify the presence of endothelial dysfunction acutely induced by the viral infection.

The secondary aim will be to evaluate the correlation between NO-mediated vascular function (evaluated by ultrasound technique) and age, anthropometric parameters (height, weight, Body Mass Index), clinical parameters, oxygenation status, physical performance and pharmacology.

The data will be analysed with the Shapiro-Wilk test to evaluate their "normality" and will be presented as mean ± standard deviation (sd) or median (interquartile range) depending on the type of distribution detected. Correlation tests (Pearson/Spearman) between ultrasound evaluation on peripheral blood flow and vessels and oxygenation levels, clinical, anthropometric and physical performance measures will then be performed. Values of p <0.05 will be considered significant.

A significant peripheral vascular dysfunction is expected to be found in post COVID individuals and to be correlated to relevant clinical variables (i.e. muscle strength, respiratory parameters, oxygenation status).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COVID-19 pneumonia
* Clinical stability condition (temperature <37.5 ° C, Respiratory Rate (RR) <22 breaths/min, Heart Rate (HR)> 50 beats/minute and <120 beats/minute, absence of major arrhythmias, hemodynamic stability)
* Possibility to reach the sitting position independently

Exclusion criteria:

-Previous cardiovascular, respiratory, neurological or orthopaedic diseases.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, from acute care hospitals, diagnosed with COVID-19 pneumonia, with documented positive throat swab, within one month from discharge.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Leg Blood Flow | Baseline
  Leg Blood Flow will be analyzed with an ultrasound examination using the Single Passive Leg Movement technique.
  In particular, the investigation consists of an ultrasound performed on the common femoral artery using Doppler method with a linear probe with a frequency of 5 MHz.
  The subject will be placed in a sitting position at rest for 20 minutes before the test is performed. The protocol consists of image acquisition for 60 seconds (basal measurement), followed by a passive flexion-extension of the knee performed by health care personnel at a rate of 1 Hz. At the end of the movement, the recording will continue for another 60 seconds.

SECONDARY OUTCOMES:
Clinical evaluations | Baseline
  Routinary measures as single anthropometric data: height (cm) and weight (Kg) and aggregate measure as body mass index (Kg/m2)
Clinical characteristics | Baseline
  Clinical course of disease (days) will be noted for all subjects
Presence of device | Baseline
  Ventilatory support (yes or no) will be noted for all subjects
Therapy | Baseline
  Drug therapy (list of drugs) will be noted for all subjects
Clinical characteristics | Baseline
  Number of comorbidities will be noted for all subjects
Biochemical evaluations - ProBNP | Baseline
  All subjects will perform blood tests to investigate bio-humoral data. Normal values: <125 pg/mL
Biochemical evaluations - D-dimer | Baseline
  All subjects will perform blood tests to investigate bio-humoral data. Normal values:<500 ng/mL FEU
Biochemical evaluations - PCR | Baseline
  All subjects will perform blood tests to investigate bio-humoral data. Normal values:<=5.00 mg/L
Functional evaluations - 1-Minute Sit To Stand | Baseline
  Therapists ask the participants to sit down on a chair without armrests. The assisted use of the arms is not allowed during the STS test. The therapists instruct the participants to complete as many sit-to-stand cycles as possible within 60 s at self-paced speed and count the number of fully-completed STS cycles. Normal values: 50/min-27/min.
Functional evaluations - 6-Minute Walking Test | Baseline
  The 6MWT is a self-paced test of walking capacity. Patients will be asked to walk as far as possible in 6 min along a flat corridor. The distance in metres is recorded. Standardised instructions and encouragement are given during the test.
  Predicted 6MW Distance follows this calculation: 361-(age in yrs x 4) + (height in cm x 2) + (HRmax/HRmax % pred x 3) - (weight in kg x 1.5) - 30 (if females).
Functional evaluations - Biceps' muscle strength with dynamometer | Baseline
  The patient will be seated with the elbow flexed 90" and forearm supinated; the dynamometer will be positioned just proximal to styloid processes and the patient will be asked to flex his elbow. Prediction equation=229.421-84.836*(0=male, 1=female) +0,165*weight-1.503*age.
Functional evaluations - Quadriceps' muscle strength with dynamometer | Baseline
  The patients will be seated with hips and knees flexed 90''; the dynamometer will be positioned just proximal to malleoli and the patient will be asked to extend his knee. Prediction equation=358.455-87.581*(0=male, 1=female) +0.297*weight-3.136*age

CONTACTS AND LOCATIONS:
Overall Officials: Mara Paneroni, PT, Principal Investigator — Istituti Clinici Scientifici Maugeri IRCCS
Locations (1):
- ICS Maugeri IRCCS, U.O. Emergenza Coronavirus di Lumezzane, Lumezzane, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guzik TJ, Mohiddin SA, Dimarco A, Patel V, Savvatis K, Marelli-Berg FM, Madhur MS, Tomaszewski M, Maffia P, D'Acquisto F, Nicklin SA, Marian AJ, Nosalski R, Murray EC, Guzik B, Berry C, Touyz RM, Kreutz R, Wang DW, Bhella D, Sagliocco O, Crea F, Thomson EC, McInnes IB. COVID-19 and the cardiovascular system: implications for risk assessment, diagnosis, and treatment options. Cardiovasc Res. 2020 Aug 1;116(10):1666-1687. doi: 10.1093/cvr/cvaa106. PMID 32352535
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Venturelli M, Layec G, Trinity J, Hart CR, Broxterman RM, Richardson RS. Single passive leg movement-induced hyperemia: a simple vascular function assessment without a chronotropic response. J Appl Physiol (1985). 2017 Jan 1;122(1):28-37. doi: 10.1152/japplphysiol.00806.2016. Epub 2016 Nov 10. PMID 27834672
- [Background] Broxterman RM, Trinity JD, Gifford JR, Kwon OS, Kithas AC, Hydren JR, Nelson AD, Morgan DE, Jessop JE, Bledsoe AD, Richardson RS. Single passive leg movement assessment of vascular function: contribution of nitric oxide. J Appl Physiol (1985). 2017 Dec 1;123(6):1468-1476. doi: 10.1152/japplphysiol.00533.2017. Epub 2017 Aug 31. PMID 28860173
- [Background] Trinity JD, Groot HJ, Layec G, Rossman MJ, Ives SJ, Runnels S, Gmelch B, Bledsoe A, Richardson RS. Nitric oxide and passive limb movement: a new approach to assess vascular function. J Physiol. 2012 Mar 15;590(6):1413-25. doi: 10.1113/jphysiol.2011.224741. Epub 2012 Feb 6. PMID 22310310
- [Background] Gifford JR, Richardson RS. CORP: Ultrasound assessment of vascular function with the passive leg movement technique. J Appl Physiol (1985). 2017 Dec 1;123(6):1708-1720. doi: 10.1152/japplphysiol.00557.2017. Epub 2017 Sep 7. PMID 28883048
- [Background] Strassmann A, Steurer-Stey C, Lana KD, Zoller M, Turk AJ, Suter P, Puhan MA. Population-based reference values for the 1-min sit-to-stand test. Int J Public Health. 2013 Dec;58(6):949-53. doi: 10.1007/s00038-013-0504-z. Epub 2013 Aug 24. PMID 23974352
- [Background] Casanova C, Celli BR, Barria P, Casas A, Cote C, de Torres JP, Jardim J, Lopez MV, Marin JM, Montes de Oca M, Pinto-Plata V, Aguirre-Jaime A; Six Minute Walk Distance Project (ALAT). The 6-min walk distance in healthy subjects: reference standards from seven countries. Eur Respir J. 2011 Jan;37(1):150-6. doi: 10.1183/09031936.00194909. Epub 2010 Jun 4. PMID 20525717
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- [Result] Paneroni M, Pasini E, Vitacca M, Scalvini S, Comini L, Pedrinolla A, Venturelli M. Altered Vascular Endothelium-Dependent Responsiveness in Frail Elderly Patients Recovering from COVID-19 Pneumonia: Preliminary Evidence. J Clin Med. 2021 Jun 9;10(12):2558. doi: 10.3390/jcm10122558. PMID 34207876